CLINICAL TRIAL: NCT06576050
Title: A Prospective Evaluation of Subjects Undergoing Weight Loss Surgery to Determine Cardiometabolic Responses to Exercise
Brief Title: WeighT LOSS Surgery and Comprehensive Cardiometabolic Responses to to EXercise
Acronym: WTLOSS-EX
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Gregory D. Lewis, M.D., Professor of Medicine, Massachusetts General Hospital
Other Study IDs: 2021P002595
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure; Obesity; Weight Loss; Heart Failure With Preserved Ejection Fraction
Keywords: heart failure; exercise capacity; obesity; weight loss; weight loss intervention
MeSH Terms: conditions — Heart Failure; Obesity; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Weight Loss Procedure: Each subject will undergo laparoscopic sleeve gastrectomy, as part of their clinical care. This is a single-arm study, in which the investigators collect data prior to the procedure, 3 months after the procedure, and 12 months after the procedure.

SUMMARY:
The goal of this study is to define how treatment of obesity impacts cardiometabolic performance during exercise in patients with established HFpEF or at risk for HFpEF. Multi-dimensional physical activity, including 6 minute walk distance, resting metabolic rate, the metabolic cost of initiating exercise, and low-level, intermediate, peak exercise, and recovery oxygen utilization patterns will be examined in relation to weight loss in people having bariatric surgery. The investigators also aim to learn more about the relationship between obesity, exercise intolerance, and heart failure with preserved ejection fraction (HFpEF). The investigators are interested in the extent to which HFpEF's manifestations are preventable or reversible with weight-loss interventions. The main questions it aims to answer are:

1. How does weight loss surgery affect comprehensive measures of physical activity?
2. What are the biochemical signatures of obesity and their reversibility in patients with HFpEF and obesity?

DETAILED DESCRIPTION:
A prospective evaluation of subjects with HFpEF or at risk for HFpEF undergoing laparoscopic sleeve gastrectomy surgery to determine cardiometabolic responses to exercise.

The investigators will prospectively evaluate twenty-one patients to determine cardiometabolic responses to exercise before and 12-months after bariatric surgery. The investigators will map pulmonary/pulmonary vascular function, ventilatory efficiency (VE/VCO2 slope); left ventricular-systemic vascular function (based on echo measures) as well as exercise blood pressure responses (SBP at 30 Watts); sympathetic nervous system function during exercise will be assessed by heart rate-O2 pulse relationships; peripheral abnormalities characteristic of HFpEF will be measured by assessment of O2 kinetics during exercise onset and recovery. Additionally, global metabolic reserve will be captured by assessment of peak VO2. The comprehensive evaluation of these patients pre- and post-weight loss will further elucidate relationships between HFpEF and obesity, and their plasticity in response to weight loss, while also setting the stage to evaluate clinical trial endpoints that influence how patients function and feel (e.g. CPET-derived exercise capacity). The investigators will also assess exercise capacity and additional markers of metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for weight loss surgery (gastric sleeve procedure)
* 40 years or older
* PMH one or more of the following:

  1. Diabetes Mellitus
  2. Hypertension requiring medical treatment
  3. Age >65 years
  4. History of HFpEF
  5. Echocardiographic findings: left atrial enlargement (LAE), left ventricular hypertrophy (LVH), or right ventricular systolic pressure >40 mmHg (RVSP)

Exclusion Criteria:

* Previous Bariatric surgery
* Pregnancy
* History of systolic heart failure, past or present LVEF of <40%
* Inability to perform exercise testing on a cycle ergometer (i.e. orthopedic conditions that preclude cycling or walking, recent systemic illness that compromises exercise capacity).
* Any contraindication to performing exercise testing or any history of ventricular arrhythmia, any recent (within the last 3 months) or untreated supraventricular arrhythmia, elevated blood pressure at the time of presentation for exercise testing (>155 mmHg systolic, or >95 mmHg diastolic blood pressure), active or recent exacerbation of congestive heart failure, or history of reactive airways disease that is induced by exercise).

  * Acute myocardial infarction (3-5 days) or unstable angina
  * Uncontrolled symptomatic arrhythmias
  * Active endocarditis
  * Acute myocarditis or pericarditis
  * Symptomatic severe aortic stenosis
  * Acute pulmonary embolism or DVT
  * Suspected dissecting aneurysm
  * Uncontrolled asthma
  * Room air desaturation to <85%
  * Acute non-cardiopulmonary disorder that may affect exercise performance (infection, orthopedic problem)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing gastric sleeve bypass weight loss procedure
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Peak VO2 | baseline to month 12
  To precisely quantify changes in peak oxygen uptake (peak VO2) achieved pre and post gastric sleeve surgery by performing cardiopulmonary exercise testing (CPET) at baseline (pre-surgery) and 12-months post-procedure (+/- 3 months). CPETs will be performed on a cycle ergometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Kenchaiah S, Evans JC, Levy D, Wilson PW, Benjamin EJ, Larson MG, Kannel WB, Vasan RS. Obesity and the risk of heart failure. N Engl J Med. 2002 Aug 1;347(5):305-13. doi: 10.1056/NEJMoa020245. PMID 12151467
- [Background] Obokata M, Reddy YNV, Pislaru SV, Melenovsky V, Borlaug BA. Evidence Supporting the Existence of a Distinct Obese Phenotype of Heart Failure With Preserved Ejection Fraction. Circulation. 2017 Jul 4;136(1):6-19. doi: 10.1161/CIRCULATIONAHA.116.026807. Epub 2017 Apr 5. PMID 28381470
- [Background] Haykowsky MJ, Nicklas BJ, Brubaker PH, Hundley WG, Brinkley TE, Upadhya B, Becton JT, Nelson MD, Chen H, Kitzman DW. Regional Adipose Distribution and its Relationship to Exercise Intolerance in Older Obese Patients Who Have Heart Failure With Preserved Ejection Fraction. JACC Heart Fail. 2018 Aug;6(8):640-649. doi: 10.1016/j.jchf.2018.06.002. Epub 2018 Jul 11. PMID 30007558
- [Background] Shah SJ, Katz DH, Selvaraj S, Burke MA, Yancy CW, Gheorghiade M, Bonow RO, Huang CC, Deo RC. Phenomapping for novel classification of heart failure with preserved ejection fraction. Circulation. 2015 Jan 20;131(3):269-79. doi: 10.1161/CIRCULATIONAHA.114.010637. Epub 2014 Nov 14. PMID 25398313
- [Background] Redfield MM, Chen HH, Borlaug BA, Semigran MJ, Lee KL, Lewis G, LeWinter MM, Rouleau JL, Bull DA, Mann DL, Deswal A, Stevenson LW, Givertz MM, Ofili EO, O'Connor CM, Felker GM, Goldsmith SR, Bart BA, McNulty SE, Ibarra JC, Lin G, Oh JK, Patel MR, Kim RJ, Tracy RP, Velazquez EJ, Anstrom KJ, Hernandez AF, Mascette AM, Braunwald E; RELAX Trial. Effect of phosphodiesterase-5 inhibition on exercise capacity and clinical status in heart failure with preserved ejection fraction: a randomized clinical trial. JAMA. 2013 Mar 27;309(12):1268-77. doi: 10.1001/jama.2013.2024. PMID 23478662
- [Background] Borlaug BA, Anstrom KJ, Lewis GD, Shah SJ, Levine JA, Koepp GA, Givertz MM, Felker GM, LeWinter MM, Mann DL, Margulies KB, Smith AL, Tang WHW, Whellan DJ, Chen HH, Davila-Roman VG, McNulty S, Desvigne-Nickens P, Hernandez AF, Braunwald E, Redfield MM; National Heart, Lung, and Blood Institute Heart Failure Clinical Research Network. Effect of Inorganic Nitrite vs Placebo on Exercise Capacity Among Patients With Heart Failure With Preserved Ejection Fraction: The INDIE-HFpEF Randomized Clinical Trial. JAMA. 2018 Nov 6;320(17):1764-1773. doi: 10.1001/jama.2018.14852. PMID 30398602
- [Background] Lewis GD, Malhotra R, Hernandez AF, McNulty SE, Smith A, Felker GM, Tang WHW, LaRue SJ, Redfield MM, Semigran MJ, Givertz MM, Van Buren P, Whellan D, Anstrom KJ, Shah MR, Desvigne-Nickens P, Butler J, Braunwald E; NHLBI Heart Failure Clinical Research Network. Effect of Oral Iron Repletion on Exercise Capacity in Patients With Heart Failure With Reduced Ejection Fraction and Iron Deficiency: The IRONOUT HF Randomized Clinical Trial. JAMA. 2017 May 16;317(19):1958-1966. doi: 10.1001/jama.2017.5427. PMID 28510680